CLINICAL TRIAL: NCT06179381
Title: FACILITY (Feeding the fAmiLy: the Intergenerational approaCh to fIght obesiTY)
Brief Title: Feeding the fAmiLy: the Intergenerational approaCh to fIght obesiTY (FACILITY)
Acronym: FACILITY
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Buzzi Children's Hospital (Other)
Collaborators: University of Pavia (Other)
Responsible Party: Principal Investigator, Valeria Calcaterra, Principal Investigator, Buzzi Children's Hospital
Other Study IDs: 02102023; CUP: F13C22001210007 (Other Grant/Funding Number: PNRR - MUR)
Record Dates: First submitted 2023-11-23; First posted 2023-12-21 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Obesity; Child Obesity; Maternal Obesity; Overweight
Keywords: Overweight; Obesity; Childhood obesity; Continuum of Care; Maternal health; Child Health; Adiposity rebound
MeSH Terms: conditions — Obesity; Pediatric Obesity; Pregnancy in Obesity; Overweight

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The FACILITY STUDY is aimed at evaluating maternal and children social, cultural, economic and lifestyle-related risk factors for the development of childhood overweight, obesity and early adiposity rebound (EAR). This study consists of two phases: a cross-sectional phase and a retrospective case-control study.

DETAILED DESCRIPTION:
The FACILITY cross-sectional study is conducted in the Buzzi Children's Hospital in Milan on children and adolescents (2-18 years old) and their mothers (≥ 18 years old). The estimated duration is 24 months.

The primary objective of the FACILITY cross-sectional is the assessment of the nutritional and socioeconomic status of mother-child dyads attending a pediatric outpatient clinic in the city of Milan, Italy (mapping). Therefore, the primary endpoint is to define the overweight and obesity prevalence in multiethnic mother-child dyads attending a pediatric outpatient clinic in the city of Milan, Italy.

The secondary objectives are: 1) Assessment of lifestyle factors and their impact on the health status of the target population. 2) Assessment of socioeconomic and cultural factors and their impact on the health status of the target population. Thus, the secondary endpoints are: 1) Impact of lifestyle on overweight and obesity in children/adolescents. 2) Impact of socio-economic-cultural factors on overweight and obesity in children/adolescents.

To mother-child dyads coming to the outpatient facilities (of the Department of Pediatrics, Buzzi Children's Hospital, Milan) and eligible in accordance with the inclusion and exclusion criteria will be proposed to participate in the study and will be given the informative material. For children and adolescents, the informed consent will be read and signed by the parents, who are the legal guardians.

On eligible subject different variables will be measured.

For mothers - Regarding lifestyle and health factors, dietary patterns will be evaluated through the Mediterranean diet (MEDI-LITE) questionnaire and through a structured interview; physical activity will be evaluated with the International Physical Activity Questionnaire (IPAQ); sleep quality will be investigated with Pittsburgh Sleep Quality Index (PSQI) questionnaire; smoking habits and alcohol consumption will be evaluated through a structured interview and anthropometric variables will include weight, height and waist circumference.

Variables referred to socio-economic and cultural factors include family relationships that will be assessed through the Child-Parent Relationship Scale - Short Form (CPRS-SF) questionnaire; the personal social capital will be investigated through the Personal Social Capital Scale (PSCS-8) questionnaire; the socio-economic status (SES) will be derived from demographic data; the neighborhood food environment characteristics, as well as the local built and social environment characteristics, will be evaluated through mapping and spatial analysis; social participation will be explored through structured interviews.

For children/adolescents - Dietary patterns will be evaluated through the Mediterranean Diet Quality Index for Children and Adolescents (KIDMED) questionnaire; physical activity will be evaluated with a structured interview for children aged 2-14 years old or with the International Physical Activity Questionnaire for Adolescents (IPAQ-A) for children aged 15-17 years old. Similarly, structured interviews will be conducted to assess sedentary screen time and sleep quality; smoking habits and alcohol consumption will be evaluated in adolescents (children aged 12-18 years old) through a structured interview and binge eating symptoms (i.e., sneaking, hiding, or hoarding food, eating in the absence of hunger) will be investigated with a structured interview. Anthropometric variables will include weight, height, adiposity rebound and waist circumference.

ELIGIBILITY:
Inclusion Criteria for mothers:

* Age ≥ 18 years old;
* Admitted to the Department of Pediatrics, Buzzi Children's Hospital, Milan, Italy;
* Written and signed informed consent.

Exclusion Criteria for mothers:

* Mother had not written and signed informed consent;
* Inability to understand the Italian and English language.

Inclusion Criteria for children:

* Age > 2 years and < 18 years old;
* Admitted to the Department of Pediatrics, Buzzi Children's Hospital, Milan, Italy;
* Mother and father/legal guardian had written and signed informed consent.

Exclusion Criteria for children:

* Endocrine disorders (hypothyroidism, hypercortisolism, growth hormone deficiency);
* Central nervous system damage (hypothalamic-pituitary damage because of surgery or trauma);
* Genetic diseases either monogenic (leptin deficiency, MC4R mutation) or pleiotropic genetic syndromes (Prader-Willi, Bardet-Biedl);
* Mother and father/legal guardian had not written and signed informed consent.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: To the patients (mother-child dyads) coming to the outpatient facilities (of the Department of Pediatrics, Buzzi Children's Hospital, Milan) and eligible in accordance with the inclusion and exclusion criteria will be proposed to participate in the study and will be given the informative material. For children and adolescents, the informed consent will be read and signed by the parents, who are the legal guardians. After the acquisition of the informed consent, the clinic information will be collected as the protocol procedure.
Sampling Method: Non-Probability Sample
Enrollment: 269 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of childhood overweight and obesity | Day 1
  Number of children with overweight or obesity divided by the total number of children.
  Diagnosis: BMI percentile in the Center for Diseases Control (CDC) growth chart (overweight: 85th-95th percentile/2-3 Z score; obesity ≥ 95th percentile/≥ 3 Z score).

SECONDARY OUTCOMES:
Mediterranean diet adherence for dyads | Day 1
  For mothers, Medi-Lite questionnaire (total score ranges between 0-18. A higher score represents higher adherence to the Mediterranean diet);
  For children, KIDMED questionnaire (total score ranges between 0-12. A higher score indicates higher adherence to the Mediterranean diet).
Dietary patterns of mothers | Day 1
  Structured interview (mother's perception of her current diet, possible dietary restrictions, traditional food/dishes consumed, influence of living in Italy on the dietary pattern).
Physical activity for dyads | Day 1
  For mothers, International Physical Activity Questionnaire short form (the questionnaire provides the total weekly Physical Activity level in metabolic equivalents (METs)/min/week; the categories are: low, moderate and vigorous physical activity).
  For children aged ≤ 14 years old: structured interview (minutes and/or hours of daily physical activity). Results will be compared with WHO guidelines.
  For children aged 15 - 17 years old, International Physical Activity Questionnaire for Adolescents (the questionnaire provides the total weekly Physical Activity level in metabolic equivalents (METs)/min/week; the categories are: low, moderate and vigorous physical activity).
Sleep quality for dyads | Day 1
  For mothers, Pittsburgh Sleep Quality Index questionnaire (total score ranges between 0-21. A higher score represents lower sleep quality).
  For children, structured interview (sleep and wake-up times, sleep regularity, average number of hours of sleep per night, difficulty falling asleep, daytime sleepiness).
Smoking habits for dyads | Day 1
  For mothers and for children aged 12 - 18 years old, structured interview: current smoking of traditional tobacco or electronic cigarettes or heated tobacco products (HTP) per day; smoking history. Based on smoking declaration, participants will be categorized as: never smoker (i.e., never smoked), past smoker (i.e., current nonsmoker), current smoke (i.e., current user of tobacco or electronic cigarette or HTP products)).
Alcohol consumption for dyads | Day 1
  For mothers and for children aged 12 - 18 years old, structured interview: current weekly alcohol consumption. Based on alcohol consumption declaration, participants will be categorized as: abstainers (i.e., subjects who do not drink alcohol, zero Units of Alcohol (U.A.)), occasional drinkers (i.e., subjects who drink less than 1 U.A./week), and daily drinkers (i.e., subjects who regularly drink alcohol, more than 1 U.A./week).
Sedentary screen time for children | Day 1
  For children, structured interview (in free time on school days: evaluation of time spent on computer, TV/movie, cell phone in leisure time on the weekend: evaluation of time spent on computer, TV/movie, cell phone).
Socio-economic status for mothers | Day 1
  For mothers: education level (none, elementary, middle school, high school, degree), nationality, profession/job, income, and housing status (owned, rented, sub-rented, social housing, guest, other, don't answer).
Family relationships for mothers | Day 1
  For mothers, Child-Parent Relationship Scale - Short Form questionnaire (higher scores indicates greater challenges in family relationships). Total score is calculated by sum. Higher total score for the closeness scale indicates higher closeness between mother and child. Higher total score for the conflict scale indicates a more conflictual relationship between mother and child.
Personal social capital for mothers | Day 1
  For mothers, Personal Social Capital Scale questionnaire (higher scores represents higher personal social capital). The summation of the two subscale (bonding capital score and bridging capital score) yield to the total social capital score. Higher total score indicates a higher social capital score.
Neighborhood food environment for mothers | Day 1
  For mothers, spatial analysis of data on location of food stores types
Social environment for mothers | Day 1
  For mothers,spatial analysis of cultural services
Social participation for mothers | Day 1
  For mothers, structured interview (activities in which the mother takes part: type and frequency of cultural, religious and recreational activities).
Weight of dyads | Day 1
  weight (kg)
Height of dyads | Day 1
  height (m)
Waist circumference of dyads | Day 1
  waist circumference (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Valeria Calcaterra, Dr, Principal Investigator — Department of Internal Medicine and Therapeutics, University of Pavia, 27100 Pavia, Italy. Pediatric Department, Buzzi Children's Hospital, 20154 Milano, Italy; Hellas Cena, Dr, Principal Investigator — Laboratory of Dietetics and Clinical Nutrition, Department of Public Health, Experimental and Forensic Medicine, University of Pavia, via Bassi 21, 27100 Pavia, Italy. Clinical nutrition Unit, General Medicine, ICS Maugeri IRCCS, 27100 Pavia, Italy

REFERENCES:
- [Derived] Vincenti A, Calcaterra V, Santero S, Viroli G, Di Napoli I, Biino G, Daconto L, Cusumano M, Zuccotti G, Cena H. FACILITY: feeding the family-the intergenerational approach to fight obesity, a cross-sectional study protocol. Front Pediatr. 2025 Mar 31;13:1450324. doi: 10.3389/fped.2025.1450324. eCollection 2025. PMID 40230801